CLINICAL TRIAL: NCT04678089
Title: Evaluating Study of Clinical Treatment of Multiple Myeloma Based on Analytical Omics
Brief Title: Evaluation of Clinical Treatment of Multiple Myeloma Based on Multi-omics
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Lihong Liu, professor, Beijing Chao Yang Hospital
Other Study IDs: 2020-9-23-7
Record Dates: First submitted 2020-11-19; First posted 2020-12-21 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma; Bortezomib
Keywords: Genomics; Metabonomics; therapeutic drug monitoring
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples and bone marrow

GROUPS / COHORTS (2):
- Health group: The healthy control group mainly collected patients with other chronic diseases or blood tumors who did not meet the exclusion criteria and were not diagnosed with multiple myeloma. Also，we need some healthy volunteers. Healthy volunteers refer to people without serious physical disease, immune disease and family history of mental illness.There is no distinction between age, gender and nationality.
- Multiple Myeloma group: In the exposure group, all patients with multiple myeloma met the inclusion and did not meet exclusion criteria, including planning for autologous stem cell transplantation or not. There is no distinction between age, gender and nationality.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Objective To observe the safety and efficacy of bortezomib related biomarkers. Including genes, metabolites, etc
  Other Names: PS-341; VELCADE
  Groups: Multiple Myeloma group

SUMMARY:
With the emergence of new drugs, the short-term survival rate of multiple myeloma has been significantly increased. However, in clinical treatment, doctors found that different patients may present different clinical efficacy and adverse reactions when using standard treatment. Some studies have shown that gene and metabolic differences in patients with multiple myeloma may be an important factor affecting clinical efficacy.

In this project, peripheral blood samples and bone marrow from patients with multiple myeloma will be studied by using the methods of genomics, proteomics, metabonomics and transcriptomics. It is expected to find biomarkers and genes related to clinical efficacy, adverse reactions, and blood concentration of bortezomib in peripheral blood samples. If the sample size is large enough, the project team expects to establish a prediction model for the efficacy and safety of bortezomib containing regimen for multiple myeloma patients through the above studies. Investigators hope that the evaluation system can provide a reference for clinical formulation of appropriate drug delivery scheme.

ELIGIBILITY:
Inclusion Criteria:

* exposure group:

  1. Patients diagnosed with multiple myeloma.
  2. Patients with fluorescence in situ hybridization report results, and try to obtain genetic diagnosis results.
* healthy control group: Patients diagnosed without multiple myeloma, such as other chronic diseases or blood tumors.

Exclusion Criteria:

1. Patients without complete clinical information.
2. Patients with malignant epidemic diseases.
3. Patients with alcohol abuse or special dietary habit .
4. Patients with digestive system diseases, such as inflammatory bowel disease, intestinal infectious disease or other diseases that may affect digestive system function.
5. Patients with a history of gastrointestinal operation.
6. Patients with severe renal insufficiency without regular dialysis.
7. Patients with other possibilities who has severe liver or kidney function injury without intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the exposure group, all patients with multiple myeloma met the inclusion and did not meet exclusion criteria, including planning for autologous stem cell transplantation or not. There is no distinction between age, gender and nationality.
  The healthy control group mainly collected patients with other chronic diseases or blood tumors who did not meet the exclusion criteria and were not diagnosed with multiple myeloma. There is no distinction between age, gender and nationality.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Treatment toxicities:neuritis | From registration to December,2022
Confirmed responses: Strictly Complete response, sCR | From registration to December,2022
Confirmed responses: Complete response, CR | From registration to December,2022
Confirmed responses: Very good partial response, VGPR | From registration to December,2022
Confirmed responses: Partial response, PR | From registration to December,2022
Confirmed responses: Minimal remission, MR | From registration to December,2022
Confirmed responses: Stable disease, SD | From registration to December,2022
Progressive disease, PD | From registration to December,2022

SECONDARY OUTCOMES:
Progression-free survival | From registration to disease progression or date of death from any cause, whichever came first, assessed up to December,2022
Overall survival | From registration to death due to any cause, assessed up to December,2022

CONTACTS AND LOCATIONS:
Overall Officials: Lihong Liu, Doctor, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijng Chao Yang Hospital, Beijing, China